CLINICAL TRIAL: NCT01643135
Title: Reduction Perioperative Bleeding in Laminectomy With Instrumentation or More Than or Equal to 3 Levels Laminectomy: The Comparison Between Placebo, and Double Doses of Tranexamic Acid (15 mg/kg and 15 mg/kg)
Brief Title: Reduction Bleeding in Laminectomy With Double Doses of Tranexamic Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Manee Raksakietisak, Associate professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: si248/2012
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Bleeding
Keywords: tranexamic acid; bleeding; blood transfusion; spine surgery
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Tranylcypromine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tranexamic acid (Active Comparator): Tranexamic acid (15 mg/kg in 0.9% NaCl and the total volume is 100 ml) will given before induction and the second dose(15 mg/kg in 0.9% NaCl and the total volume is 100 ml) will be given at 3 hours after the first dose.
  Interventions: Drug: tranexamic acid
- 0.9% NaCl (Placebo Comparator): 0.9% NaCl 100 ml will be given as a placebo before induction and 3 hours after the first dose
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: tranexamic acid — Transamine acts as antifibrinolysis which looks alike 0.9% NaCl (placebo)
  Other Names: transamine (Daiichi-Sankyo, Japan)
  Arms: tranexamic acid
Drug: 0.9% NaCl — 0.9% NaCL (NSS) is clear fluid which looks alike tranexamic acid
  Other Names: NSS
  Arms: 0.9% NaCl

SUMMARY:
Tranexamic acid has benn widely used to reduce perioperative bleeding in several operations such as cardiac surgery, liver transplant and joint arthroplasty with good results. Few studies in laminectomy had conflicting results and varying in doses. The objective is to compare perioperative bleeding in major laminectomy between patients receive doubles doses of tranexamic acids (15 mg/kg and 15 mg/kg) with who receive pacebo (0.9% NaCl).

DETAILED DESCRIPTION:
78 patients undergoing major laminectomy (with instrumentation or equal or more than 3 levels laminectomy) will be enrolled. We exclude patients who age over 65, anemia, allergy to tranexamic acid, history of deep vein thormbosis (DVT), ischemic heart disease (IHD), pulmonary embolism (PE), strokes, liver disease, chronic kidney disease with creatinine >2.0 mg/dl, and coagulopathy. After randomization, before induction and 3 hour after the first dose, patients will receive study drug or placebo intravenously. The standard anesthesia and monitoring will be tha same for all of the patients. Perioperative mild hypotensive technique will be used with the mean arterial pressure more than 60 mmHg and nearly the end, the blood pressure will be back to normal for the bleeding check. Hematocrit will be monitored at the begining and every two hours. Blood will be given if the hematocrit is below 30%. The perioperative fluid will be managed by anesthesiologist who will not know the patients' groups. The next morning, the hematocrit and blood creatinine will be checked and if the hematocrit is lower than 30%, blood will be given. Perioperative blood loss, total fluid and blood transfusion within 24 hours will be recorded. If there are any suspected symptoms and signs of DVT, angina, CHF, PE, strokes or other complications, the necessory investigations will be done for the definite dignosis and the appropriate treatment will be started immediately.

ELIGIBILITY:
Inclusion Criteria:

* has laminectomy with instrumentation or equal or more than 3 levels laminectomy
* age 18-65 years
* ASA 1-3
* elective operation

Exclusion Criteria:

* allergy to tranexamic acid
* anemia (Hb<12 g/dl in female or Hb<13 g/dl in male)
* history of CVT, IHD, PE, strokes
* liver disease
* chronic kidney disease with creatinie>2.0 mg/dl
* receive anticoagulant or coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
perioperative blood loss | 24 hours
  Intraoperative and postoperative blood loss will be measured by from swab, suction and vaccum drainage

SECONDARY OUTCOMES:
perioperative blood transfusion | 24 hours
  When the blood loss more than acceptable and the hematocrit below 30%, the packed red cell will be given.

CONTACTS AND LOCATIONS:
Overall Officials: Manee Raksakietisak, MD, Principal Investigator — Mahidol University
Locations (1):
- Manee Raksakietisak, Bangkok, Thailand